CLINICAL TRIAL: NCT04506385
Title: Effects of Probiotics Administration on Human Metabolic Phenotype
Brief Title: Metabolomic Effects of Probiotics Administration
Acronym: MAPPINg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probiotical S.p.A. (Industry)
Collaborators: University of Florence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 294/CE
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Metabolomic Profile
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A - L. delbrueckii LDD01 probiotic bacterial strain administered in sachets of 2 grams (Active Comparator): L. delbrueckii LDD01 probiotic bacterial strain
  Interventions: Dietary Supplement: probiotics
- B - Bifidobacterium longum DLBL probiotic bacterial strain administered in sachets of 2 grams (Active Comparator): Bifidobacterium longum DLBL probiotic bacterial strain
  Interventions: Dietary Supplement: probiotics
- C - LP01, LF16, LR06 and B. longum 04 administered in sachets of 2 grams (Active Comparator): L. plantarum LP01, L.fermentum LF16, L. rhamnosus LR06 and B. longum 04: low dosage; probiotic bacterial strains blend
  Interventions: Dietary Supplement: probiotics
- D - LP01, LF16, LR06 and B. longum 04 administered in sachets of 2 grams (Active Comparator): L. plantarum LP01, L.fermentum LF16, L. rhamnosus LR06 and B. longum BL04: high dosage; probiotic bacterial strains blend
  Interventions: Dietary Supplement: probiotics

INTERVENTIONS:
Dietary Supplement: probiotics — In the first phase: 10 subjects have added in the diet a daily dose of 1 billion of freeze-dried LDD01 probiotics (A arm), 12 individuals are supplemented with a daily dose of 1 billion of the DLBL mix (B arm). In the second phase: 10 individuals are supplemented with a daily low dose of probiotics blend (C arm) and 10 individuals are supplemented with a daily high dose of probiotics blend (D arm).

SUMMARY:
Background: The establishment of the beneficial interactions between the host and its microbiota is essential for the development and correct functioning of the organism, since microflora alterations can lead to many chronic degenerative diseases. In this context, probiotics are used to improve balanced microbial communities and therefore exert substantial health-promoting effects to the host.

Objective: The aim of the present study is to monitor the molecular outcomes, obtained by gut microflora modulation through probiotic treatment, on human urine and serum metabolic profiles, with a 1H-Nuclear Magnetic Resonance -based metabolomic approach.

DETAILED DESCRIPTION:
Design: In a first phase twenty-two healthy subjects are enrolled in the study and administered with Lactobacillus delbrueckii subs. delbrueckii and/or a mix of 5 biotypes of Bifidobacterium longum for 8 weeks. In the second phase subjects are enrolled in the study and administered with Lactobacillus rhamnosus, Lactobacillus plantarum, Lactobacillus fermentum and Bifidobacterium longum at two different concentration. During the course of the study all the probiotic types were administered both singularly and in combination. From each subject urine and serum samples are collected before and during the supplementation and are analysed by nuclear magnetic resonance spectroscopy and statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

- healthy subjects

Exclusion Criteria:

* previous surgery on the intestinal tract;
* a probiotic / prebiotic and antibiotic treatments within 3 and 1 months, respectively, before the beginning of the study;
* subjects have changed drastically their diet or lifestyle during the study.

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
metabolomic profile | 20 days
  To monitor the molecular outcomes, obtained by gut microflora modulation through probiotic treatment, on human urine and serum metabolic profiles, with a 1H-Nuclear Magnetic Resonance-based metabolomic approach

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera-Universitaria Maggiore della carità di Novara, Novara, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No